CLINICAL TRIAL: NCT05523362
Title: Feasibility and Clinical Utility of the Dexcom G6 Continuous Glucose Monitoring Device for the Care of Patients With Type 2 Diabetes Not Using Insulin Therapy
Brief Title: Feasibility and Clinical Utility of the Dexcom G6 Continuous Glucose Monitoring Device for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ian J. Neeland, MD (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ian J. Neeland, MD, Director, UH Center for Cardiovascular Prevention, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20221148
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: The device is used in blinded mode where both patient and provider are blinded to the data only during Phase 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Blinded followed by Unblinded (Experimental): During Phase 1 (10 days), the patient wears the Dexcom G6 Pro CGM in blinded mode and is unaware and unable to access the data. The patient performs standard care, self-monitoring with twice daily glucose checks using standard finger-sticks and a glucometer device. During this phase, the medical providers are also blinded to the CGM data and continue standard care without any specific intervention.
  During Phase 2 (3 months), the patient wears the Dexcom G6 Personal CGM in un-blinded mode and the medical providers have access to the data via Clarity and/or direct download via the transmitter. CGM data are collected continuously in each phase and at the end of each phase.
  Interventions: Device: Dexcom continuous glucose monitor

INTERVENTIONS:
Device: Dexcom continuous glucose monitor — The investigational device used in this study is the Dexcom G6 Pro/Personal Continuous Blood Glucose Monitoring system.

SUMMARY:
The objective of this study is to evaluate the feasibility and clinical utility of a continuous glucose monitoring device (CGM, Dexcom G6) for the care of patients with type 2 diabetes who are on non-insulin therapies.

DETAILED DESCRIPTION:
The investigational device used in this study is the Dexcom G6 Pro/Personal Continuous Blood Glucose Monitoring system.

This investigation is a 2-phase sequential study with patients serving as their own controls. The demographics, medical history, anthropometric and laboratory data are collected at baseline for each patient. During Phase 1 (10 days), the patient wears the Dexcom G6 Pro CGM in blinded mode and is unaware and unable to access the data. The patient performs standard care, self-monitoring with twice daily glucose checks using standard finger-sticks and a glucometer device. During this phase, the medical providers are also blinded to the CGM data and continue standard care without any specific intervention.

During Phase 2 (3 months), the patient wears the Dexcom G6 Personal CGM in un-blinded mode and the medical providers have access to the data via Clarity and/or direct download via the transmitter. CGM data are collected continuously in each phase and at the end of each phase. Anthropometric and laboratory data (including HB A1c) are collected. Medical providers are also un-blinded and adjust medical recommendations and interventions, in part based on CGM data, as appropriate.

All patients will receive usual care which will include individual and virtual lifestyle education, virtual support group, M.D. visits, medication interventions, referrals to support programs outside the scope of CINEMA program and nursing support

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes of any duration
* Hb A1c ≥ 7% (no upper limit)
* BMI ≥ 30 kg/m2
* Ability to wear CGM (e.g. no dermatological issue precluding device insertion)
* Access to a smartphone device

Exclusion Criteria:

* Any insulin use in the past 3 months
* Planned use of insulin in the next 6 months
* Presence of a blood disorder (such as sickle cell anemia) making glycosylated hemoglobin measurement inaccurate
* Current use of a weight loss medication
* Unable or uncomfortable with wearing a CGM device

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Neeland, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 people did not meet eligibility criteria. They were consented but did not participate in the study. A total of 56 participants signed consents and only 47 fully completed both phases of the study.
Groups:
- Dexcom G6 Continuous Glucose Monitoring Device: During Phase 1 (10 days), the patient wears the Dexcom G6 Pro CGM in blinded mode and is unaware and unable to access the data. The patient performs standard care, self-monitoring with twice daily glucose checks using standard finger-sticks and a glucometer device. During this phase, the medical providers are also blinded to the CGM data and continue standard care without any specific intervention.
  During Phase 2 (3 months), the patient wears the Dexcom G6 Personal CGM in un-blinded mode and the medical providers have access to the data via Clarity and/or direct download via the transmitter. CGM data are collected continuously in each phase and at the end of each phase.
Period: Phase 1- Blinded (10 Days)
Arm/Group | Dexcom G6 Continuous Glucose Monitoring Device
Started | 56
Completed | 47
Not Completed | 9
Not completed — Unable to contact | 2
Not completed — High stress, did not want to continue | 1
Not completed — Technical issues with device | 4
Not completed — did not meet eligibility criteria | 2
Period: Phase 2- Unblinded (3 Months)
Arm/Group | Dexcom G6 Continuous Glucose Monitoring Device
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 2 people did not meet eligibility criteria. They were consented but did not participate in the study. A total of 56 participants signed consents and only 47 fully completed both phases of the study.
Groups:
- Blinded Followed by Unblinded: During Phase 1 (10 days), the patient wears the Dexcom G6 Pro CGM in blinded mode and is unaware and unable to access the data. The patient performs standard care, self-monitoring with twice daily glucose checks using standard finger-sticks and a glucometer device. During this phase, the medical providers are also blinded to the CGM data and continue standard care without any specific intervention.
  During Phase 2 (3 months), the patient wears the Dexcom G6 Personal CGM in un-blinded mode and the medical providers have access to the data via Clarity and/or direct download via the transmitter. CGM data are collected continuously in each phase and at the end of each phase.
  Dexcom continuous glucose monitor: The investigational device used in this study is the Dexcom G6 Pro/Personal Continuous Blood Glucose Monitoring system.
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 32
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Glucose Levels as Measured by Continuous Glucose Monitor
Description: Average glucose on CGM
Time Frame: 0, 30, 60, 90 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mg/dl
  Day 0 | 184 (55.7)
  Day 30 | 148.6 (45.4)
  Day 60 | 144.8 (45.3)
  Day 90 | 147.2 (44.7)

2. Primary Outcome: Change in Time in Range as Measured by Continuous Glucose Monitor
Description: Time in range is the time spent in the acceptable glucose range between 80-180 mg/dl. This time in range is noted as a proportion of time that the blood glucose is in this range out of the total time. So if the person's glucose is in this range 70% of the time (and out of it 30%), then Time in Range is 70%.
Time Frame: 0, 30, 60, 90 days
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
percentage of time in range
  Day 0 | 57.8 (32.5)
  Day 30 | 82 (22.7)
  Day 60 | 83.8 (23.8)
  Day 90 | 82.5 (24.6)

3. Primary Outcome: Change in Glucose Variability as Measured by Continuous Glucose Monitor
Description: Glucose variability on CGM is defined as standard deviation of the all recorded glucose values.
Time Frame: 0, 30, 60, 90 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mg/dl
  Day 0 | 26.2 (8.9)
  Day 30 | 24.1 (7.5)
  Day 60 | 24.1 (7.7)
  Day 90 | 24 (6.6)

4. Secondary Outcome: Change in Hemoglobin A1c From Blood Test
Description: Glycosylated hemoglobin
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated hemoglobin
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
percentage of Glycosylated hemoglobin
  Day 0 | 8.4 (1.8)
  Day 90 | 6.9 (1.2)

5. Secondary Outcome: Change in Total Cholesterol From Blood Test
Description: Total cholesterol
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mg/dl
  Day 0 | 162.6 (45.6)
  Day 90 | 143.6 (45.2)

6. Secondary Outcome: Change in Low Density Lipoprotein Cholesterol From Blood Test
Description: LDL-C
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mg/dl
  Day 0 | 82.8 (37)
  Day 90 | 73.6 (38.5)

7. Secondary Outcome: Change in High Density Lipoprotein Cholesterol From Blood Test
Description: HDL-C
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mg/dl
  Day 0 | 45.5 (12.4)
  Day 90 | 43.9 (10.5)

8. Secondary Outcome: Change in Triglycerides From Blood Test
Description: Triglycerides
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mg/dl
  Day 0 | 173.3 (110.4)
  Day 90 | 131.2 (69.7)

9. Secondary Outcome: Change in Body Mass Index From Height and Weight
Description: BMI
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
kg/m2
  Day 0 | 37.7 (6.1)
  Day 90 | 34.9 (5.9)

10. Secondary Outcome: Change in Systolic Blood Pressure From Automated Cuff
Description: Systolic blood pressure
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mmHg
  Day 0 | 134.8 (16.3)
  Day 90 | 126.0 (15.2)

11. Secondary Outcome: Change in Diastolic Blood Pressure From Automated Cuff
Description: Diastolic blood pressure
Time Frame: 0 and 90 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
mmHg
  Day 0 | 79.4 (6.7)
  Day 90 | 75.8 (7.3)

12. Secondary Outcome: Picture Your Plate Dietary Assessment Questionnaire
Description: Picture Your PlateTM is a brief (48-question) dietary assessment questionnaire developed to assess how well an individual's eating habits align with current evidence-based recommendations. Picture Your Plate provides a total score ranging from 0 to 96, with a higher score indicating healthier food choice awareness.
Time Frame: 0, 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
score on a scale
  Day 0 | 61 (12.4)
  Day 90 | 65.5 (17.7)

13. Secondary Outcome: Type 2 Diabetes Distress Screening Scale (T2-DDAS)
Description: The T2-DDAS is a self-report survey that has 29 items. Each item rated on a 1 to 5 scale:
  Mean score < 2.0 indicate little or no distress.
  Mean score between 2.0 and 2.9 indicate moderate distress.
  Mean score > 3.0 indicate high distress
Time Frame: 0, 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
score on a scale
  Day 0 | 2.4 (0.9)
  Day 90 | 1.6 (0.5)

14. Secondary Outcome: International Physical Activity Questionnaire (IPAQ)
Description: The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. This measure assesses the types of intensity of physical activity that people do as part of their daily lives. The estimate is measured as total physical activity in MET-min/week. Lower scores mean less total amount and intensity of physical activity and higher scores mean greater total amount and intensity of physical activity in a given week.
Time Frame: 0, 90 days
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 47
minutes per week
  Day 0 | 2864.8 (3329)
  Day 90 | 3445.4 (3040)

15. Secondary Outcome: Glucose Monitoring Satisfaction Survey
Description: The GMSS is a reliable, valid measure of glucose device satisfaction in its T1D form and in its insulin-using T2D form. It provides a comprehensive profile of sources of device satisfaction for use in clinical care and research.
Time Frame: 90 days
Population: No data was collected.
Arm/Group | Blinded Followed by Unblinded
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Baseline through end of the Unblinded Phase, approximately 100 days
Description: 2 people did not meet eligibility criteria. They were consented but did not participate in the study. A total of 56 participants signed consents and only 47 fully completed both phases of the study.
Groups:
- Blinded: During Phase 1 (10 days), the patient wears the Dexcom G6 Pro CGM in blinded mode and is unaware and unable to access the data. The patient performs standard care, self-monitoring with twice daily glucose checks using standard finger-sticks and a glucometer device. During this phase, the medical providers are also blinded to the CGM data and continue standard care without any specific intervention.
- Unblinded: During Phase 2 (3 months), the patient wears the Dexcom G6 Personal CGM in un-blinded mode and the medical providers have access to the data via Clarity and/or direct download via the transmitter. CGM data are collected continuously in each phase and at the end of each phase.
Arm/Group | Blinded | Unblinded
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/47
Other Adverse Events (participants affected / at risk) | 0/56 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT05523362/Prot_SAP_000.pdf